CLINICAL TRIAL: NCT04903678
Title: Intrathecal Chemotherapy for Central Nervous System Metastasis in Retinoblastoma (A Multicenter Prospective Single Arm Trial)
Brief Title: Intrathecal Chemotherapy for Central Nervous System Metastasis in Retinoblastoma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Eye & ENT Hospital of Fudan University (Other)
Collaborators: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other); Children's Hospital of Fudan University (Other)
Responsible Party: Principal Investigator, Jiang Qian, Professor, Eye & ENT Hospital of Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FD-EENT-2021056
Record Dates: First submitted 2021-05-22; First posted 2021-05-26 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Retinoblastoma, Extraocular
Keywords: retinoblastoma; central metastases; intrathecal Chemotherapy
MeSH Terms: conditions — Retinoblastoma | interventions — Melphalan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- intrathecal chemotherapy in patients with central metastases (Experimental): Systemic chemotherapy and intrathecal chemotherapy are performed every 3 weeks. After three treatment cycles, the treatment response is comprehensively evaluated including cerebrospinal fluid, intracranial and orbital tumors. If necessary, local radiotherapy and arterial interventional chemotherapy are performed for local solid tumors. Cerebrospinal fluid is detected in each treatment cycle. If RB tumor cells still exist in cerebrospinal fluid, chemotherapy and intrathecal chemotherapy are continued until the end event. If cerebrospinal fluid was negative, intrathecal chemotherapy is supplemented for another 2 cycles with a total of 6 cycles of systemic chemotherapy. The patients are followed up after treatment.
  Interventions: Drug: Melphalan

INTERVENTIONS:
Drug: Melphalan — Melphalan is performed for intrathecal chemotherapy

SUMMARY:
Retinoblastoma is the most common intraocular malignancy in infancy and childhood. The overall survival rate of retinoblastoma was reported to exceed 95% when children were early diagnosed with localized intraocular phase. The advanced retinoblastoma cases with central nervous system metastasis (CNS)is associated with exceedingly poor prognosis. CNS metastasis is the main cause of death in retinoblastoma. Meningeal involvement combined with spinal cord membrane involvement might be due to the meninges invasion and/or the spreading of CSF.

As the most sensitive drug to retinoblastoma tumor cells in vitro, melphalan is the most important drug in the local treatment of retinoblastoma, and it is also an irreplaceable drug in the current eye preservation treatment, which greatly improves the success rate of eye preservation for advanced retinoblastoma. According to the research and the practice of vitreous injection (melphalan), the drug concentration in vitreous can effectively kill retinoblastoma tumor cells.

It is reasonable to speculate that the tumor cells in CSF can be effectively killed by melphalan. Therefore, based on the above background, this study will explore the effectiveness and feasibility of intrathecal injection of melphalan in patients with CNS metastasis of retinoblastoma through a multicenter prospective study.

ELIGIBILITY:
Inclusion Criteria:

* The pathological diagnosis was retinoblastoma. According to the IRSs (International retinoblastoma staging system) staging system, the stage was IVB
* CSF tumor cells on cytology, or radiographic evidence of NM on MRI scans and histologic diagnosis of systemic malignancy needed
* KPS≥60%
* Adequate bone marrow and organ function
* The parents signed the informed consent and were willing to accept the treatment and follow-up.

Exclusion Criteria:

* 1.Eye diseases other than retinoblastoma
* The eyes were infected within 30 days before screening
* There was a history of surgery and / or unhealed wound within 1 month before enrollment .
* Those who have allergic reaction or allergic history to chemotherapeutic drugs.
* Infectious diseases requiring oral, intramuscular or intravenous administration.
* Patients with systemic immune diseases.
* Active disseminated intravascular coagulation.
* Abnormal coagulation function.
* Abnormal bone marrow and organ function.
* Uncontrollable clinical problems.
* The researchers believe that those who need to be excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2028-05-01 (Estimated); Study Completion 2030-05-01 (Estimated)

PRIMARY OUTCOMES:
progression-free survival | 1 year
  living subjects
overall survival at 2-year interval | 2 years
  living subjects
overall survival at 5-year interval | 5 years
  living subjects
response rate | 1 year
  tumor-free subjects
disease-free survival at 2-year interval | 2 years
  tumor-free subjects
disease-free survival at 5-year interval | 5 years
  tumor-free subjects

SECONDARY OUTCOMES:
Number of Participants with Arachnoiditis | 2 years
  A disorder characterized by inflammation of the arachnoid membrane and adjacent subarachnoid space.
Number of Participants with Encephalopathy | 5 years
  A disorder characterized by a pathologic process involving the brain.
Number of Participants with Headache | 2 years
  A disorder characterized by a sensation of marked discomfort in various parts of the head, not confined to the area of distribution of any nerve.
Number of Participants with Encephalomyelitis infection | 1 year
  A disorder characterized by an infectious process involving the brain and spinal cord tissues.
Health-Related Quality of life | 10 years
  The health-related quality of life will be assessed based on the EORTC (European Organisation for Research and Treatment of Cancer) Quality of Life Questionnaire Core 30 (QLQ-C30) downloaded from https://www.eortc.org. This 30-item questionnaire includes five functional scales, three symptom scales, a global health status / QoL scale, and six single items. The multi-item scales include a different set of items. Each item includes four subscales, namely "Not at all" (1 point), "A little" (2 points), "Quite a bit" (3 points) and "Very much" (4 points)
Ophthalmic Cancer-Related Quality of life | 10 years
  The ophthalmic cancer-related quality of life will be assessed based on the EORTC (European Organisation for Research and Treatment of Cancer) Quality of Life Questionnaire Ophthalmic Cancer Module 30 (QLQ-OPT30)
  - Page 4 of 6 [DRAFT] - downloaded from https://www.eortc.org. The QLQ-OPT30 comprises of 30 questions assessing vision impairment (9 items), functional problems due to vision impairment (8 items), eye symptoms (6 items), worry about recurrent disease (2 items), problems with appearance (1 items), problems driving (2 items), headache (1 item), problems reading (1 item). Each item includes four subscales, namely "Not at all" (1 point), "A little" (2 points), "Quite a bit" (3 points) and "Very much" (4 points).

CONTACTS AND LOCATIONS:
Overall Officials: Jiang Qian, MD, Principal Investigator — Fudan Eye & ENT Hospital
Locations (1):
- Fudan Eye & ENT Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code